CLINICAL TRIAL: NCT02149498
Title: Mapping Functional Networks of Brain Activity (Brain Network Activation, BNA) Based on Analysis of Evoked Response Potential (ERP) Signals for Healthy Controls Evoked Response Potential (ERP) Signals for Healthy Controls and Patients With Parkinson Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dr. Oren Cohen (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Oren Cohen, MD, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Other Study IDs: PD-MAG-01
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson; EEG; BNA
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Parkinson Disease (PD): Idiopathic PD patients (according to the UK PD Society brain bank clinical diagnostic criteria (bradykinesia plus at least one other cardinal feature of PD, no atypical features or secondary cause)
- Healthy Controls: Healthy individuals

SUMMARY:
A cornerstone in PD research is the investigation of neurophysiological changes as potential biomarkers that could help in tracking disease progression and response to therapies. Electroencephalography (EEG) could provide a non-invasive and relatively cheap tool for identification of such biomarkers. In this study we will use high-density electroencephalograph (EEG) recording, in order to develop a platform of biomarkers that could be more sensitive and reliable to disease progression and response to therapeutic intervention than standard clinical measures.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic PD patients (according to the UK PD Society brain bank clinical diagnostic criteria (bradykinesia plus at least one other cardinal feature of PD, no atypical features or secondary cause) and HC aged 40-80 years
2. PD patients Hoehn and Yahr stages I to IVStable PD therapy

Exclusion Criteria:

* In the investigator's opinion, any unstable or clinically significant condition that would impair the participants' ability to comply with study requirements.
* Patients or HC with significant psychiatric symptoms or history
* BDI score <14
* MMSE <25
* Treatment with neuroleptics.
* For PD patients: Hoehn and Yahr Stage 5
* PD Patients with severe dyskinesia or tremor
* PD Patients with atypical Parkinsonism or secondary Parkinsonism
* History or evidence of neurological problems: cerebrovascular disease, previous head injury or neurosurgical interventions.
* Currently with lice or open wounds on scalp.
* Significant sensory deficits, e.g., deafness or blindness
* Current drug abuse or alcoholism.
* Pregnancy or not using a reliable method of birth control.
* Participation in current clinical study or clinical study within 30 days prior to this study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 patients with idiopathic Parkinson's disease (PD) 50 Healthy controls (HC)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Functional networks of brain activity in Idiopathic PD patients and healthy individuals measured using analysis of EEG Event Related Potential | 2 WEEKS
  The study outcome measure are functional networks of brain activity of PD patients and healthy individuals established based on an analysis of EEG data recorded while study subjects perform ERP tasks

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Hassin, Dr., Study Director — Sheba Medical Center; Oren Cohen, Dr., Principal Investigator — Sheba Medical Center